CLINICAL TRIAL: NCT02970968
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Assess the Efficacy of VLY-686 (Tradipitant) in Relieving Symptoms of Gastroparesis
Brief Title: Study to Assess the Efficacy of VLY-686 in Relieving Symptoms of Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VP-VLY-686-2301
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — LY686017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Drug (Experimental): VLY-686 (Tradipitant) oral capsule for 4 weeks.
  Interventions: Drug: VLY-686 (Tradipitant)
- Placebo (Placebo Comparator): Placebo oral capsule for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VLY-686 (Tradipitant) — oral capsule
  Arms: Study Drug
Other: Placebo — placebo oral
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to be conducted in the United States. One hundred fifty (150) subjects diagnosed with gastroparesis, who satisfy the selection criteria for the study, will be randomized to one of two treatment groups, active or placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to be conducted in the United States. One hundred fifty (150) subjects diagnosed with gastroparesis, who satisfy the selection criteria for the study, will be randomized to one of two treatment groups, active or placebo.

The study is divided into two phases: the screening phase and the evaluation phase. The screening phase includes a screening visit to evaluate subjects' preliminary eligibility for the study. During the screening phase, subjects will collect diary data for at least 4 weeks. The evaluation phase includes 4 weeks of randomized double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with gastroparesis;
2. Subjects must agree to the use of contraception
3. Ability and acceptance to provide written informed consent;
4. Willing to participate in the pharmacogenomics sample collection;
5. Willing and able to comply with all study requirements and restrictions
6. Willing to not participate in any other interventional trial for the duration of their participation.

Exclusion Criteria:

1. Another active disorder or treatment which could explain or contribute to symptoms in the opinion of the Investigator (including but not limited to gastric malignancy, neurological disorder, or heavy doses of strong anticholinergics);
2. Pregnancy or nursing;
3. History of intolerance and/or hypersensitivity to medications similar to VLY-686 (Tradipitant) and its accompanying excipients;
4. Use of another NK1 antagonist or palonosetron;
5. Exposure to any investigational medication, including placebo, within 60 days of the Baseline Visit;
6. Any other reason as determined by the Investigator which may lead to an unfavorable risk-benefit of study participation, may interfere with study compliance, or may confound study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Vanda Investigational Site, Dothan, Alabama
  - Vanda Investigational Site, Huntsville, Alabama
  - Vanda Investigational Site, Tucson, Arizona
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Chula Vista, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, Palo Alto, California
  - Vanda Investigational Site, San Francisco, California
  - Vanda Investigational Site, Jacksonville, Florida
  - Vanda Investigational Site, Largo, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Athens, Georgia
  - Vanda Investigational Site, Elgin, Illinois
  - Vanda Investigational Site, Indianapolis, Indiana
  - Vanda Investigational Site, Louisville, Kentucky
  - Vanda Investigational Site, Marrero, Louisiana
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, Wyoming, Michigan
  - Vanda Investigational Site, Minneapolis, Minnesota
  - Vanda Investigational Site, Pascagoula, Mississippi
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Great Neck, New York
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Raleigh, North Carolina
  - Vanda Investigational Site, Salisbury, North Carolina
  - Vanda Investigational Site, Huber Heights, Ohio
  - Vanda Investigational Site, Mentor, Ohio
  - Vanda Investigational Site, Tulsa, Oklahoma
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Chattanooga, Tennessee
  - Vanda Investigational Site, Jackson, Tennessee
  - Vanda Investigational Site, Nashville, Tennessee
  - Vanda Investigational Site, El Paso, Texas
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Richardson, Texas
  - Vanda Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlin JL, Lieberman VR, Dahal A, Keefe MS, Xiao C, Birznieks G, Abell TL, Lembo A, Parkman HP, Polymeropoulos MH. Efficacy and Safety of Tradipitant in Patients With Diabetic and Idiopathic Gastroparesis in a Randomized, Placebo-Controlled Trial. Gastroenterology. 2021 Jan;160(1):76-87.e4. doi: 10.1053/j.gastro.2020.07.029. Epub 2020 Jul 18. PMID 32693185

RESULTS

PARTICIPANT FLOW:
Groups:
- Tradipitant: oral, 85 mg/day given bid
- Placebo: oral, matching placebo given bid
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 77 | 75
Completed | 72 | 68
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.16) | 46.4 (13.46) | 45.9 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 66 | 65 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease Etiology [Count of Participants; unit: Participants]
  Idiopathic | 46 | 45 | 91
  Diabetic | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Nausea Severity
Description: The Gastroparesis Core Symptom Daily Diary (GCSDD) is a patient reported diary that asks patients to rate the worst occurrence of each cardinal symptom of gastroparesis (nausea severity, early satiety, postprandial fullness, bloating, and abdominal pain) in the past 24 hours on a Likert scale from 0 (no symptoms) to 5 (very severe). Change from baseline in average nausea severity score is calculated as the weekly average post value minus baseline value of the daily nausea severity score from the GCSDD. A negative change indicates improvement.
Time Frame: 4 weeks
Population: The ITT Population included any subject randomized into the study who received a dose of study medication and had at least 1 valid postbaseline efficacy measurement while on study medication. The ITT Population comprised 141 subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
score on a scale (change from baseline) | -1.25 [-1.53 to -0.98] | -0.73 [-1.02 to -0.44]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0099, Mixed Models Analysis

2. Secondary Outcome: Weekly % Nausea-Free Days
Description: The Gastroparesis Core Symptom Daily Diary (GCSDD) is a patient reported diary that asks patients if they have had any nausea over the past 24 hours and if yes, to rate the worst occurrence in the past 24 hours on a Likert scale from 1 (very mild) to 5 (very severe). Change in weekly percentage of nausea-free days from baseline is calculated as weekly average post value minus baseline value. Baseline is defined as the average of all nonmissing values in the screening phase (4 weeks).
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage (%) of nausea-free days
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
Percentage (%) of nausea-free days | 28.81 [21.09 to 36.53] | 15.00 [6.94 to 23.07]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0160, Mixed Models Analysis

3. Secondary Outcome: Daily Average Vomiting Frequency, Change From Baseline
Description: The Gastroparesis Core Symptom Daily Diary (GCSDD) is a patient reported diary that asks patients if they have vomited in the past 24 hours and how many times they vomited in the past 24 hours. Change from baseline in the weekly average of daily vomiting frequency is calculated as the weekly average post value minus baseline value of the daily daily vomiting frequency from the GCSDD. Baseline is defined as the average of all non-missing values in the screening phase (4 weeks). A negative change indicates improvement.
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: weekly average of daily vomit episodes
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
weekly average of daily vomit episodes | -0.49 [-0.64 to -0.34] | -0.26 [-0.42 to -0.10]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .039, Mixed Models Analysis

4. Secondary Outcome: Gastroparesis Cardinal Symptom Index (GCSI), Change From Baseline
Description: The GCSI is a subject reported outcome administered in-clinic with a 2-week recall period to measure the severity of symptoms in gastroparesis. The GCSI is composed of 9 items based on three subscales: post-prandial fullness/early satiety (4 items); nausea/vomiting (3 items), and bloating (2 items). The severity of each symptom is rated on a six-point Likert response scale. The minimal scale value = 0 (none) and the maximum scale value = 5 (very severe). GCSI Total score is constructed as the average of the three symptom sub-scales. Higher score is indicative of greater symptom severity.
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
score on a scale (change from baseline) | -0.93 [-1.14 to -0.73] | -0.58 [-0.80 to -0.36]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0223, Mixed Models Analysis

5. Secondary Outcome: PAGI-SYM, Change From Baseline
Description: The PAGI-SYM is a patient reported outcome which asks patients to describe the severity of their symptoms over the last two weeks to measure symptom severity for gastroparesis, functional dyspepsia, and gastroesophageal reflux disease. The measure consists of 20 symptom severity items, which cover the following domains: nausea/vomiting, fullness/early satiety, bloating, upper abdominal pain, heartburn/regurgitation, and lower abdominal pain. This questionnaire includes the Gastroparesis Cardinal Symptom Index (GCSI). The severity of each symptom is rated on a six-point Likert response scale. The minimal scale value = 0 (none) and the maximum scale value= 5 (very severe). PAGI-SYM Total score is constructed as the average of the six symptom sub-scales and a higher score is indicative of greater symptom severity.
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
score on a scale (change from baseline) | -0.93 [-1.12 to -0.74] | -0.65 [-0.86 to -0.45]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0497, Mixed Models Analysis

6. Secondary Outcome: CGI-S, Change From Baseline
Description: The Clinician Global Impression of Severity (CGI-S) is a 7-point scale on which the clinician rates the severity of the patient's gastroparesis at the time of the assessment and refers to the degree of illness at the time of the visit and during the 2 weeks before the visit. The CGI-S is rated on the following 7-point scale: 1: normal, not at all ill; 2: borderline ill: 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; 7: among the most extremely ill patients. Change from baseline is calculated as post value minus baseline value. A negative change indicates improvement.
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
score on a scale (change from baseline) | -1.13 [-1.36 to -0.91] | -0.74 [-0.98 to -0.50]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0207, Mixed Models Analysis

7. Secondary Outcome: PGI-C
Description: The Patient Global Impression of Change (PGI-C) is a patient reported questionnaire with a 7-point rating scale where the participant rates his/her own improvement in overall symptoms relative to the baseline assessment. Is is rated as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Higher scores indicate a worse outcome.
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
score on a scale (change from baseline) | 2.66 [2.40 to 2.93] | 3.06 [2.78 to 3.35]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0429, Mixed Models Analysis

8. Post Hoc Outcome: Change From Baseline in Average Nausea Severity; Baseline Vomiting Group
Description: as for outcome 1
Time Frame: 4 weeks
Population: The baseline vomiting group subpopulation was defined as all subjects who reported at least 1 episode of vomiting during the screening period and consisted of 101 of 141 (72%) patients of the ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
score on a scale (change from baseline) | -1.43 [-1.72 to -1.14] | -0.42 [-0.76 to -0.07]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p < .0001, Mixed Models Analysis

9. Post Hoc Outcome: GCSDD, % Nausea-Free Days; Baseline Vomiting Group
Description: The Gastroparesis Core Symptom Daily Diary (GCSDD) is a patient reported diary that asks patients to rate the worst occurrence of each cardinal symptom of gastroparesis in the past 24 hours on a scale from 0 (no symptoms) to 5 (very severe).
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage (%) of nausea-free days
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
Percentage (%) of nausea-free days | 32.3 [23.8 to 40.8] | 7.6 [-2.3 to 17.5]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0003, Mixed Models Analysis

10. Post Hoc Outcome: GCSDD, Daily Average Vomiting Frequency, Change From Baseline; Baseline Vomiting Group
Description: The Gastroparesis Core Symptom Daily Diary (GCSDD) is a patient reported diary that asks patients to rate the worst occurrence of each cardinal symptom of gastroparesis in the past 24 hours on a scale from 0 (no symptoms) to 5 (very severe). Change from baseline is calculated as post value minus baseline value. A negative change indicates improvement.
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: weekly average of daily vomit episodes
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
weekly average of daily vomit episodes | -0.69 [-0.89 to -0.49] | -0.32 [-0.56 to -0.08]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .023, Mixed Models Analysis

11. Post Hoc Outcome: Gastroparesis Cardinal Symptom Index (GCSI), Change From Baseline; Baseline Vomiting Group
Description: as for outcome 4
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
score on a scale (change from baseline) | -1.10 [-1.33 to -0.87] | -0.60 [-0.88 to -0.32]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0078, Mixed Models Analysis

12. Post Hoc Outcome: PAGI-SYM, Change From Baseline; Baseline Vomiting Group
Description: as for outcome 5
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
score on a scale (change from baseline) | -1.06 [-1.28 to -0.85] | -0.69 [-0.95 to -0.43]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0294, Mixed Models Analysis

13. Post Hoc Outcome: CGI-S, Change From Baseline; Baseline Vomiting Group
Description: The Clinician Global Impression of Severity (CGI-S) is a 7-point scale on which the clinician rates the severity of the patient's gastroparesis at the time of the assessment and refers to the degree of illness at the time of the visit and during the 2 weeks before the visit. The CGI-S is rates on the following 7-point scale: 1: normal, not at all ill; 2: borderline ill: 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; 7: among the most extremely ill patients. Change from baseline is calculated as post value minus baseline value. A negative change indicates improvement.
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
score on a scale (change from baseline) | -1.24 [-1.49 to -0.99] | -0.79 [-1.08 to -0.49]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0229, Mixed Models Analysis

14. Post Hoc Outcome: PGI-C; Baseline Vomiting Group
Description: as for outcome 7
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (change from baseline)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
score on a scale (change from baseline) | 2.52 [2.24 to 2.81] | 3.24 [2.90 to 3.59]
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0018, Mixed Models Analysis

15. Post Hoc Outcome: Nausea Responder Rate (%)
Description: Defined as a nausea score of very mild or better (≤1) in average daily nausea severity at week 4. Nausea severity is rated on a Likert scale from 0 (none) to 5 (very severe).
Time Frame: 4 weeks
Measure: Number; unit: Percentage (%) of nausea responders
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
Percentage (%) of nausea responders | 32.9 | 11.8
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0013, Mixed Models Analysis

16. Post Hoc Outcome: Nausea Responder Rate (%); Baseline Vomiting Group
Description: as for outcome 15
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Number; unit: Percentage (%) of nausea responders
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
Percentage (%) of nausea responders | 36.2 | 6.9
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0001, Mixed Models Analysis

17. Post Hoc Outcome: Complete Nausea Responder Rate (%)
Description: Defined as a nausea score of 0 in at week 4. Nausea severity is rated on a Likert scale from 0 (none) to 5 (very severe).
Time Frame: 4 weeks
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
Percentage (%) of participants | 15.07 | 4.4
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .018, Mixed Models Analysis

18. Post Hoc Outcome: Complete Nausea Responder Rate (%); Baseline Vomiting Group
Description: Defined as a nausea score of 0 at week 4. Nausea severity is rated on a Likert scale from 0 (none) to 5 (very severe).
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
Percentage (%) of participants | 17.24 | 4.65
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0164, Mixed Models Analysis

19. Post Hoc Outcome: Percentage of Participants With Clinically Meaningful Improvement on Total GCSI Score
Description: Defined as 1-point or greater improvement on their GCSI total score from baseline to week 4. The GCSI is a subject reported outcome. Part I consists of the traditional GCSI and severity rating of upper abdominal pain and severity of overall symptoms on a 0 (none) to 5 (very severe) Likert scale. Part II uses a 7-point rating scale for the subject to rate their own improvement relative to baseline. Symptoms are rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. The GCSI subscale scores, nausea/vomiting (3 items), postprandial fullness/early satiety (4 items), bloating (2 items), and upper abdominal pain (2 items), are calculated by taking the mean of non-missing items in each subscale; the subscale scores vary from 0 (none or absent) to 5 (very severe). The total score is calculated by taking the mean of the three subscales (except upper abdominal pain and overall symptom item).
Time Frame: 4 weeks
Measure: Number; unit: Percentage (%)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 73 | 68
Percentage (%) | 46.6 | 23.5
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0053, Mixed Models Analysis

20. Post Hoc Outcome: Percentage of Participants With Clinically Meaningful Improvement on Total GCSI Score; Baseline Vomiting Group
Description: as for outcome 19
Time Frame: 4 weeks
Population: as for outcome 8
Measure: Number; unit: Percentage (%)
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 58 | 43
Percentage (%) | 51.7 | 23.3
Statistical Analysis 1: Comparison: Tradipitant vs Placebo; Test type: Superiority; p = .0020, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All safety analyses are based on the safety population.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/75
Other Adverse Events (participants affected / at risk) | 31/77 | 20/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant (N=77) | Placebo (N=75)
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant (N=77) | Placebo (N=75)
Diarrhea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 3
Somnolence (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Fatigue (General disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Studies are needed to determine the mechanisms by which tradipitant reduces nausea and vomiting, and powered to assess idiopathic and diabetic gastroparesis separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02970968/Prot_SAP_000.pdf